## **MEMORANDUM**

## Department of Veterans Affairs

<name> VA Medical Center

| Medical Cent | er Director | Date |
|---|---|---|
| Point of Con<br><name> VA N</name> | tact<br>/ledical Center | Date |
| This documer | nt should be kept on file at both institutions. | |
| | ing below also agree to provide relevant site-spec<br>as outlined in the site preparation checklist. | ific information to the Function |
| With respect to acknowledge Function QU Durham IRB of Associate Exercisearch open program-relative participation is | to the individual research project specified above to that the <a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href="research"><a href<="" td=""><th>arch by implementing the ne attached memo from the ified by Barbara Hyduke, MSA, I Care (10P4G) to be a non-will participate in clinical VAMC will participate in any ion activities, employee</th></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a></a> | arch by implementing the ne attached memo from the ified by Barbara Hyduke, MSA, I Care (10P4G) to be a non-will participate in clinical VAMC will participate in any ion activities, employee |
| Name of Inst | itution Providing IRB Review: Durham VAMC | |
| <b>Principal Inv</b><br>Van Houtven, | estigator(s): Susan N. Hastings, MD, MHS ( <u>susa</u><br>PhD; Kelli Allen, PhD (coordinating site: Durham | n.hastings@va.gov); Courtney<br>VA) |
| Name of Res<br>2.0") | earch Project: Optimizing Function and Independ | dence QUERI ("Function QUER |
| To: | <name> VA Medical Center</name> | |
| Subject: | Participation Agreement for the Function QUERI | STRIDE Project |
| From: | Susan N. Hastings, MD, MHS | |
| Date: | July 20, 2022 | |